CLINICAL TRIAL: NCT04374097
Title: Level and Predictors of Trauma-symptoms Among Health Workers and Public Service Providers During the COVID-19 Outbreak
Status: Completed | Type: Observational
Sponsor: University of Oslo (Other)
Collaborators: Modum Bad (Other)
Responsible Party: Principal Investigator, Sverre Urnes Johnson, Associate Professer Sverre Urnes Johnson, University of Oslo
Other Study IDs: REK125510(2)
Record Dates: First submitted 2020-05-02; First posted 2020-05-05 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Post Traumatic Stress Disorder; Anxiety; Depression
Keywords: COVID-19; Health personnel; Predictor; PTSD; Anxiety; Depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the levels of trauma and mental symptoms (i.e., depression and anxiety) among health workers and public service providers during the strict social distancing government-initiated non-pharmacological interventions (NPI's) related to the COVID-19 pandemic. The study also aims to investigate predictors of trauma-symptoms.

DETAILED DESCRIPTION:
Hypotheses/Research questions:

H1: Health employees and public service providers working directly with COVID-19 will have higher PTSD-symptoms, anxiety, depression and health anxiety, compared to health workers and public service providers working indirectly with the virus.

H2: Presence of a psychological disorder, anxiety and depression will predict PTSD symptoms. Those reporting having a diagnosis will reveal higher PTSD-symptoms. Higher levels of anxiety and depression will be associated with higher PTSD-symptoms.

H3: Emotional support, burnout, health-anxiety, worry about job and economy, interpersonal problems and metacognition will predict PTSD-symptoms controlling for direct vs. indirect exposure to trauma, psychological diagnosis, demographic variables (age and gender, living with a partner, living with children, anxiety and depression. Higher level of burnout, health-anxiety, worry about job and economy, interpersonal problems and metacognition will be associated with higher PTSD-symptoms. Higher emotional support will be associated with lower PTSD-symptoms.

Participants were asked to fill out a set of validated questionnaires including demographic variables, psychological symptoms and PTSD-symptoms. Some questionnaires are given as a whole, whereas other questions includes theoretically-driven selections of items from validated questionnaires. This study is part of a 'The Norwegian COVID-19, Mental Health and Adherence project". The study involves a Cross-sectional survey design. Health personnel and public service providers where systematically targeted through various channels: e.g., primarily through systematically reaching out to all hospitals in Norway and inviting health personnel to participants, through contacting the Associations of all major health-worker groups (i.e., Norwegian Medical Doctors Association; Norwegian Nurses Association, Norwegian Psychologists Association; and other associations related to health-workers) through national TV, national, regional and local radio stations, and national, regional and local newspapers in the different regions of the country, as well as Facebook groups in the different regions of the country. Additionally, a random selection of those qualifying as health-care workers were randomly targeted on Facebook by a Facebook Business algorithm. Public service providers were recruited trough Facebook. Politicians where also systematically contacted, with all political parties being contacted and subsequently sending an e-mail with the survey to their members.

Data collection started during the time-period with the strictest and equal number of government-initiated non-pharmacological interventions (NPI's) in Norway, and data collection was stopped once these NPI's were modified or new information about NPI's were added. The data include one directly identifiable variable (contact information) for participants in accordance to the General Data Protection Regulation (GDPR) law in EU, which is to give the participants the opportunity to have their data deleted upon request. Data are thus kept on a safe server belonging to the University of Oslo and is accessed first following de-identification. The project outline and study plan was also registered upon application to the Norwegian "Regional Ethical Committee" 10 days before data collection, a committee which evaluate the rational for data collection and hypotheses as well as evaluate the ethical aspects of the study before allowing the data to be collected.

Measures

PCL-5, PHQ-9; GAD-7; demographic variables (gender; age; relationship/marital status; living with children and number of children; employment status; education level); situational variables related to Covid-19, worry about own health and worry about economy/work, emotional support, interpersonal problems, burnout, metacognitions and whether one has a psychological diagnosis or not. The outcome variable is PCL-5. Predictors are specified in the hypothesis-section.

Indices:

Given Acceptable Cronbach's alpha (above 0.7) the investigators combined four items that measure health anxiety and fear of death related to COVID-19. Furthermore two items will be combined to represent worry about work and economy. Two items on emotional support were combined. On the CAS1 four items were combined into the subscale "positive metacognition" and four items were combined into the subscale "negative metacognition". Interpersonal problems consisted of 13 items selected from the IIP-64. Burnout was measured with a single item

Inference:

Given the large sample size in this study, the investigators pre-defined our significance level:

p < 0.01 to determine significance

Sample size 'Norwegian COVID-19 and Mental Health and Adherence Project' involves multiple studies, where some involve a Complex Systems (Network analysis approach). These multivariate analyses require large samples and power analysis was conducted accordingly. Following power analysis guidelines by Fried & Cramer (2017), it is recommended that the number of participants be at the very least three times larger than the number of estimated parameters. However, more conservative recommendations by Roscoe (1975) for multivariate research, recommends sample size that is ten times larger than the number of estimated parameters. Thus, with the more conservative estimates by Roscoe, an optimal sample size included 1900.

Statistical models:

Descriptive statistics with frequency tables including N, mean and SDs or median and interquartile range depending on the data will be presented. A cut-off of 31 on the PCL-5 will be used together with the DSM-5 diagnostic guidelines applied to the PCL-5 to categorize participants as fulfilling the PTSD symptom criteria or not. Participants indicating scores of 2 or above on at least one of five re-experiencing symptoms, one of two avoidance symptoms, two of seven symptoms of negative alterations in cognition and mood and two of six arousal symptoms were classified as fulfilling the PTSD symptom criteria. Subclinical PTSD will be assessed by specifying how large part of the sample which fulfil parts of the PTSD-criterias. The results will be benchmarked against national and international studies.

Independent sample t-tests or Mann-Whitney U tests, depending on level of skewness, will be used to compare the PCl-5 scores of those working direct vs. indirect with COVID-19 patients. A One-way ANOVA or Kruskal-Wallis test, depending on level of skewness, will be conducted to exploratory investigate differences between the different types of health-workers (e.g. medical doctor and clinical psychologists) and public service providers (e.g., politicians, social security). If there is significant differences between the groups the investigators will either use a post hoc test, Tukey (HSD) or Dunn-Bonferroni, depending on wether a parametric or non-parametric test has been used.

Two multiple regression analyses will be conducted with PCL-5 as the dependent variable. Specific predictors of the different regression are listed in the hypothesis section. Multicollinearity and other assumptions will be checked; if the multicollinearity assumption is violated (if VIF > 5 and Tolerance < 0.2.

Exploratory analyses:

Exploratory: Examine the differences in levels of trauma, anxiety, depression and health anxiety among different health workers, public service providers and demographic subgroups.

The investigators may also do other exploratory analysis that not yet thought of at the time of pre-registration. Such analysis will be explicitly stated as exploratory.

Note that this project outline, study plan and analysis was registered upon application to the Regional Committees for Medical and Health Research Ethics (REC) and Norwegian Centre for Research Data.

ELIGIBILITY:
Inclusion Criteria:

- All health-care or public service provides above 18 was eligible for inclusion in this study. Vulnerable health-care or public service providers was in this sample defined as doctors, nurses, psychologists, and any other health-care workers, as well as politicians and social workers. The participants reported if they worked directly or indirectly with COVID-19 patients.

Given the time-sensitivity of the project and the strict and time-consuming process of getting approval to access registry data, the investigators did not apply for access to registry data (e.g., address, phone or e-mails of the general population), as such data access is highly strict and regulated in Norway and the time-frame of such an application could have encompassed variation in an important variable the investigators wished to hold constant (namely identifical NPIs (non-pharmacological interventions) employed over the time-frame of data collection). Thus, the investigators did not apply for registry data, but still attempted to obtain a probability sample through the means elaborated below.

Health personnel and public service providers where systematically targeted through various channels: e.g., primarily through systematically reaching out to all hospitals in Norway and inviting health personell to participants, through contacting the Associations of all major health-worker groups (i.e., Norwegian Medical Doctors Association; Norwegian Nurses Association, Norwegian Psychologists Association; and other associations related to health-workers) through national TV, national, regional and local radio stations, and national, regional and local newspapers in the different regions of the country, as well as Facebook groups in the different regions of the country. Additionally, a random selection of those qualifying as health-care workers were randomly targeted on Facebook by a Facebook Business algorithm. Public service providers were recruited trough Facebook. Politicians where also systematically contacted, with all political parties being contacted and subsequently sending an e-mail with the survey to their members.

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Both Biological Sex and self-representation of gender are measured. All participants are welcome to partake in the study.
Study Population: Eligible participants are health-care or public service provides above 18 in Norway.
  To hold the NPI variable constant, the stopping rule of data collection was at once if the NPIs were modified; new NPI were added; NPIs were removed; or novel information about modification of NPIs were given.
Sampling Method: Probability Sample
Enrollment: 1778 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-04-07 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | All data was collected between March 31st 2020 and April 7th 2020, a period where the NPIs (nonpharmacological interventions) against the COVID-19 pandemic were identical and constant in Norway
  PCL-5 is 20-item self-administered questionnaire which assesses the full domain of the DSM-5 PTSD diagnosis. The self-report rating scale is 0-4 for each symptom. Rating scale descriptors are: "Not at all," "A little bit," Moderately," "Quite a bit," and "Extremely."The PCL-5 has four subscales, corresponding to each of the symptom clusters in the DSM-5.

SECONDARY OUTCOMES:
Patient Health Questionnaire 9 (PHQ-9) | All data was collected between March 31st 2020 and April 7th 2020, a period where the NPIs (nonpharmacological interventions) against the COVID-19 pandemic were identical and constant in Norway
  The Patient Health Questionnaire 9 (PHQ-9; Kroenke, Spitzer & Williams, 2001) is used to measure symptoms of depression in accordance with the diagnostic criteria for major depressive disorder. The questionnaire consists of nine items where each is scored on a four-point Likert scale (0-3), with the range of scores from 0 to 27.
The Generalized Anxiety Disorder 7 (GAD-7) | All data was collected between March 31st 2020 and April 7th 2020, a period where the NPIs (nonpharmacological interventions) against the COVID-19 pandemic were identical and constant in Norway]
  The Generalized Anxiety Disorder 7 (GAD-7; Spitzer, Kroenke, Williams & Löwe, 2006) is a questionnaire consisting of seven items measuring symptoms of anxiety and worry. The items are scored on a four-point Likert scale (0-3), with the scores ranging from 0 to 21.
Health anxiety | All data was collected between March 31st 2020 and April 7th 2020, a period where the NPIs (nonpharmacological interventions) against the COVID-19 pandemic were identical and constant in Norway
  Symptoms of health anxiety was measured with two items from the validated Health Anxiety Inventory (HAI), one item measuring specific fear of being infected by coronavirus, and an item measuring fear of dying by the coronavirus. All items used a Likert scale from 0-3, and the new total score of health anxiety had a range from 0-12.

CONTACTS AND LOCATIONS:
Overall Officials: Sverre Urnes Johnson, PhD, Principal Investigator — University of Oslo & Modum Bad; Omid Ebrahimi, Principal Investigator — University of Oslo & Modum Bad; Asle Hoffart, PhD, Principal Investigator — Modum Bad & University of Oslo
Locations (1):
- University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No